CLINICAL TRIAL: NCT00791843
Title: The Effect of GHRH Therapy on Myocardial Structure and Function in Congestive Heart Failure
Acronym: GHRH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Grant AG00599; PP1:MGH 2004p-000099
Record Dates: First submitted 2008-11-13; First posted 2008-11-17 (Estimated); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Congestive Heart Failure
Keywords: CHF
MeSH Terms: conditions — Heart Failure | interventions — Growth Hormone-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GHRH and placebo (Experimental): Everyone will receive 12 weeks of GHRH and 12 weeks of Placebo
  Interventions: Drug: Growth hormone releasing hormone/ placebo

INTERVENTIONS:
Drug: Growth hormone releasing hormone/ placebo — 12 weeks of drug at max dose of 2mg/day administered in 4 pulses at 11pm, 1am, 3am, and 5am, followed by 6 weeks of washout period, then 12 weeks of placebo or vise versa- 12 weeks of placebo, 6 weeks washout, 12 weeks of drug.

SUMMARY:
PP1- The purpose of this study is to determine whether giving more of the hormone produced by everyone called growth hormone releasing hormone (GHRH) can improve heart function in individuals with congestive heart failure. You must be 50 years old or older, have a diagnosis of congestive heart failure, and have a high likelihood of having lower than normal growth hormone effect. GHRH is approved by the US FDA for treatment in children with growth hormone deficiency because GHRH stimulates Growth Hormone (GH). Its use for treatment of congestive heart failure in adults is investigational.

Growth hormone releasing hormone is a hormone produced in the brain. We will be using synthetic hormone made in the laboratory. It is identical to the hormone in the brain.

Many older people, due to aging have low levels of growth hormone. The aim of this study is to find out whether restoring growth hormone levels to the levels found in younger individuals and then maintaining those levels for 12 weeks will help strengthen heard muscles in older persons with congestive heart failure.

DETAILED DESCRIPTION:
PP1- The overall purpose of this study is to evaluate the effects of Growth Hormone Releasing Hormone (GHRH) on cardiac structure and function in subjects aged 50 years and older with a diagnosis of congestive heart failure in a single blinded (to the subject) randomized treatment/placebo study design. They will receive 12 weeks of drug or placebo, 6 weeks of washout, and 12 weeks of placebo or drug- whichever they didn't receive in the first 12 weeks. The hypotheses are: 1)normal aging is associated with evidence of declining somatotrophic activity exemplified by IGF-1 levels; 2) GHRH can raise levels of Growth hormone and IGF-1 in elderly individuals in a dose dependent fashion with minimal deleterious side effects; 3) GHRH will produce measurable increments in myocardial performance and structure and demonstrated growth of peripheral musculature; 4) the combination of these benefits will result in better quality of life due to the improvement of overall cardiac function.

ELIGIBILITY:
INCLUSION CRITERIA:

* subjects will be at least 50 years of age,
* women who are post-menopausal.
* clinical evidence of congestive heart failure, with ongoing management by conventional medical therapy
* a left ventricular ejection fraction below 40% as measured by echocardiogram performed within 6 months of study enrollment.
* Left ventricular end-diastolic dimension greater than 60 mm as measured by an echocardiogram performed within 6 months of study enrollment.
* regular heart rate/pacer
* hemodynamically stable and able to complete symptom-limited bicycle ergometry exercise test;
* and be in New York Heart Association Classification II or III.

EXCLUSION CRITERIA:

* Subjects with hematocrit equal to or less than 33%;
* body mass index equal to or greater than 40;
* unstable angina within six months;
* inducible ischemia by exercise stress testing, radionuclide scintigraphy, or dobutamine echocardiography;
* known or suspected myocarditis;
* known or suspected restrictive or infiltrative cardiomyopathy;
* coronary artery stenosis >70% and < 100% by catheterization should such data be available;
* inadequate cardiac echo window;
* primary diastolic dysfunction in heart failure
* inability to perform cycle ergometry;
* critical aortic stenosis;
* severe mitral regurgitation by Doppler echocardiography;
* uncontrolled or poorly controlled hypertension;
* hypertrophic cardiomyopathy;
* renal failure, determined by creatinine > 2.0.
* untreated thyroid disease;
* active alcoholism,
* breast cancer;
* prostate cancer;
* inability to provide informed consent;
* uncontrolled hyperlipidemia; (Triglycerides >1200 and/or LDL > 160)
* patients with known bleeding disorders;
* patients using atropine, artane, scopolamine, and cogentin.
* Subjects who have implanted devices that contain metal and are not adherent to the body will be excluded from the MRI testing in this study. These devices include pacemakers, implanted ICD's, infusion pumps, nerve stimulators, metal debris in the eye, or loose metal, such as shrapnel or a bullet.
* Inability to lie flat on back for an extended period of time. The MRI testing requires this posture.
* History of any noncutaneous malignancy within 5 years of screening.

STUDY TERMINATION CRITERIA:

The following clinical events will define drop-points for worsening clinical conditions and will terminate subject involvement in the study:

* Unstable angina
* Acute myocardial infarction (chest pain with EKG changes and increased troponin)
* NYHA Class IV heart failure for greater than one week (a brief episode of NYHA Class IV heart failure may result from medical or dietary indiscretion, adverse effects of non-study medications, poorly controlled hypertension and other potentially reversible mechanisms)
* Documented sustained ventricular tachycardia
* Resuscitated cardiac arrest
* Unexplained syncope
* Diagnosis of sleep apnea that is not medically supervised.
* Symptomatic documented bradycardia
* Diagnosis of a new non-cutaneous malignancy
* Developing exclusion criteria
* Stroke
* Death

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital/ Geriatric Research, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Period: Overall Study
Arm/Group | GHRH and Placebo
Started | 0 (Data unavailable for the study)
Completed | 0 (Data unavailable for the study)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Arm/Group | GHRH and Placebo
Number analyzed (Participants) | 0
Age, Categorical — Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Sex: Female, Male — Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: PP1- Serum IGF-1 Levels, DXA, Resting Metabolic Rate, Total Body Water, 3-D Echo, Cardiac MRI, Dobutamine Stress Echocardiogram, Ergometry, General Health Assessment, Physical Exam
Time Frame: baseline, 12, 18, and 30 weeks
Population: Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Arm/Group | GHRH and Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Description: Data unavailable for study, PI is deceased and all staff associated with study have left the institution.
Arm/Group | GHRH and Placebo
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Data unavailable for study, PI is deceased and all staff associated with study have left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes